CLINICAL TRIAL: NCT01472562
Title: Phase II Study of Lenalidomide Plus Rituximab in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: Lenalidomide Plus Rituxan for Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1103011566
Record Dates: First submitted 2011-03-24; First posted 2011-11-16 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mantle Cell Lymphoma
Keywords: mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients (Experimental): Induction Phase (week 1 - 48):
  * Lenalidomide will be given at 20 mg/day for days 1-21 of a 28-day cycle for 12 cycles. If no excess toxicity is observed the dose will be increased to 25 mg/day.
  * Rituximab will be administered at 375 mg/m2 per dose for a total of 9 doses. The first 4 doses will be administered weekly starting on day 1 of lenalidomide (e.g. days 1, 8, 15 and 22). Subsequent rituximab doses will be administered for one dose each at weeks 12, 20, 28, 36 and 44.
  Maintenance Phase (week 49 - progression of disease):
  * Lenalidomide will be given at 15 mg/day for days 1-21 of a 28-day cycle.
  * Rituximab at 375 mg/m2 per dose will be administered for one dose every 8 weeks, starting at week 52.
  Interventions: Drug: lenalidomide; Biological: rituximab

INTERVENTIONS:
Drug: lenalidomide — Induction phase: 20 mg/day for days 1-21 of a 28-day cycle for 12 cycles. If no excess toxicity is observed the dose will be increased to 25 mg/day.
  Maintenance phase: Lenalidomide will be given at 15 mg/day for days 1-21 of a 28-day cycle.
  Other Names: revlimid
Biological: rituximab — Induction phase: Rituximab will be administered at 375 mg/m2 per dose for a total of 9 doses. The first 4 doses will be administered weekly starting on day 1 of lenalidomide (e.g. days 1, 8, 15 and 22). Subsequent rituximab doses will be administered for one dose each at weeks 12, 20, 28, 36 and 44.
  Maintenance phase: Rituximab at 375 mg/m2 per dose will be administered for one dose every 8 weeks, starting at week 52.
  Other Names: rituxan

SUMMARY:
This is a phase II, multicenter study to determine the efficacy and safety of first-line lenalidomide plus rituximab therapy in patients with mantle cell lymphoma who have received no prior systemic therapy.

DETAILED DESCRIPTION:
Induction Phase (week 1 - 48):

* Lenalidomide will be given at 20 mg/day for days 1-21 of a 28-day cycle for 12 cycles. If no excess toxicity is observed the dose will be increased to 25 mg/day.
* Rituximab will be administered at 375 mg/m2 per dose for a total of 9 doses. The first 4 doses will be administered weekly starting on day 1 of lenalidomide (e.g. days 1, 8, 15 and 22). Subsequent rituximab doses will be administered for one dose each at weeks 12, 20, 28, 36 and 44.

Maintenance Phase (week 49 - progression of disease):

* Lenalidomide will be given at 15 mg/day for days 1-21 of a 28-day cycle.
* Rituximab at 375 mg/m2 per dose will be administered for one dose every 8 weeks, starting at week 52.

Response Assessment

* Year 1-2: Conventional restaging CT scan (or MRI) with IV contrast every 3 months from cycle 1 day 1 of the study.
* Year 3 onwards: Conventional restaging CT scan (or MRI) with IV contrast every 6 months until progression.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age > = 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Histologically confirmed diagnosis of mantle cell Non-Hodgkin's Lymphoma with cyclin D1 overexpression by immunohistochemistry, and a characteristic immunophenotypic profile with CD5(+), CD23(-), CD20(+), and CD10(-). In tumor tissues with negative cyclin D1, evidence of cyclin D2 or D3 overexpression by immunohistochemistry will be acceptable.
* No prior systemic therapy for lymphoma including chemotherapy or immunotherapy. Patients may have received involved-field radiation therapy which has been discontinued at least 4 weeks prior to treatment in this study.
* Patient has measurable disease as defined by a tumor mass > 1.5 cm in one dimension.
* Low and intermediate-risk disease as defined by MIPI score.
* Subject who the investigator considers that chemotherapy is not indicated.
* ECOG performance status of < = 2 at study entry.
* Laboratory test results within these ranges:

  * Absolute neutrophil count > = 1000 /mm³
  * Platelet count > = 75,000 /mm³
  * Calculated creatinine clearance ≥ 30 ml/min by Cockcroft-Gault formula • Total bilirubin < = 2 x ULN
  * AST (SGOT) and ALT (SGPT) < = 3 x ULN.
* Disease free of prior malignancies for > = 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or localized prostate cancer.
* All subjects must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Subjects of reproductive potential agree to use birth control throughout their participation in this study, and for three months following study termination.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days). FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
* Asymptomatic carriers of hepatitis B virus can be considered for study if they agree to and comply with close monitoring and suppressive therapy with lamivudine during treatment and for additional six months after coming off study.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Patient on corticosteroids within two weeks prior to study entry, except for prednisone < = 10 mg/day or equivalent for purposes other than treating MCL.
* Known hypersensitivity to thalidomide.
* Any prior use of lenalidomide.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Known central nervous system (CNS) involvement by lymphoma.
* Patient at high risk for deep vein thrombosis not willing to take DVT prophylaxis.
* Patient has had major surgery within the last 3 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-07-29 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Ruan, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Weill Cornell Medical College, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Yamshon S, Chen GZ, Gribbin C, Christos P, Shah B, Schuster SJ, Smith SM, Svoboda J, Furman RR, Leonard JP, Martin P, Ruan J. Nine-year follow-up of lenalidomide plus rituximab as initial treatment for mantle cell lymphoma. Blood Adv. 2023 Nov 14;7(21):6579-6588. doi: 10.1182/bloodadvances.2023010606. PMID 37682791
- [Derived] Ruan J, Martin P, Christos P, Cerchietti L, Tam W, Shah B, Schuster SJ, Rodriguez A, Hyman D, Calvo-Vidal MN, Smith SM, Svoboda J, Furman RR, Coleman M, Leonard JP. Five-year follow-up of lenalidomide plus rituximab as initial treatment of mantle cell lymphoma. Blood. 2018 Nov 8;132(19):2016-2025. doi: 10.1182/blood-2018-07-859769. Epub 2018 Sep 4. PMID 30181173
- [Derived] Ruan J, Martin P, Shah B, Schuster SJ, Smith SM, Furman RR, Christos P, Rodriguez A, Svoboda J, Lewis J, Katz O, Coleman M, Leonard JP. Lenalidomide plus Rituximab as Initial Treatment for Mantle-Cell Lymphoma. N Engl J Med. 2015 Nov 5;373(19):1835-44. doi: 10.1056/NEJMoa1505237. PMID 26535512
- See also: HemOnc clinical trials listing at Weill Cornell Medical College — http://www.cornellmedicine.org/trials/cancer-and-blood-disorders/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Study Treatment Arm
Period: Induction Phase (Week 1- 48)
Arm/Group | All Patients
Started | 38
Completed | 27
Not Completed | 11
Period: Maintenance Phase (Week 49 to PD)
Arm/Group | All Patients
Started | 27
Completed | 4
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 65 [42 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The primary endpoint of overall response rate will be estimated and a 95% confidence interval will be estimated via binomial proportions.
Time Frame: 30 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | All Patients
Number analyzed (Participants) | 33
percentage of patients | 92 [78 to 98]

2. Secondary Outcome: Number of Participants With Progression-free Survival
Description: Secondary endpoints of progression-free survival (PFS), overall survival (OS), and time to the next treatment will be assessed by Kaplan-Meier survival analysis.PFS will be defined as the time from the first treatment day until objective or symptomatic progression or death. The outcome measure is the number of participants who achieved PFS.
Time Frame: 10 years
Population: We enrolled a total of 38 patients (all evaluable for safety), but only 36 were evaluable for responses. Two patients could not be evaluated because they had an inflammatory syndrome ("tumor flare") during the first cycle and were withdrawn before response assessment.
Measure: Number; unit: participants
Groups:
- All Patients: Induction Phase (week 1 - 48):
  * Lenalidomide will be given at 20 mg/day for days 1-21 of a 28-day cycle for 12 cycles. If no excess toxicity is observed the dose will be increased to 25 mg/day.
  * Rituximab will be administered at 375 mg/m2 per dose for a total of 9 doses. The first 4 doses will be administered weekly starting on day 1 of lenalidomide (e.g. days 1, 8, 15 and 22). Subsequent rituximab doses will be administered for one dose each at weeks 12, 20, 28, 36 and 44.
  Maintenance Phase (week 49 - progression of disease):
  * Lenalidomide will be given at 15 mg/day for days 1-21 of a 28-day cycle.
  * Rituximab at 375 mg/m2 per dose will be administered for one dose every 8 weeks, starting at week 52.
  lenalidomide: Induction phase: 20 mg/day for days 1-21 of a 28-day cycle for 12 cycles. If no excess toxicity is observed the dose will be increased to 25 mg/day.
  Maintenance phase: Lenalidomide will be given at 15 mg/day for days 1-21 of a 28-day cycle.
  rituximab: Induction phase: Rituximab will be administered at 375 mg/m2 per dose for a total of 9 doses. The first 4 doses will be administered weekly starting on day 1 of lenalidomide (e.g. days 1, 8, 15 and 22). Subsequent rituximab doses will be administered for one dose each at weeks 12, 20, 28, 36 and 44.
  Maintenance phase: Rituximab at 375 mg/m2 per dose will be administered for one dose every 8 weeks, starting at week 52.
Arm/Group | All Patients
Number analyzed (Participants) | 36
participants | 21

3. Secondary Outcome: Number of Participants With Overall Survival
Description: Secondary endpoints of progression-free survival (PFS), overall survival (OS), and time to next treatment will be assessed by Kaplan-Meier survival analysis. Overall survival will be defined as the time from first treatment day until death.
  The outcome measures is the number of participants who achieved OS.
Time Frame: 10 years
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 36
participants | 24

4. Secondary Outcome: Time to Next Treatment
Description: Median amount of time (in months) from start of study treatment to next treatment
Time Frame: 10 years
Population: Data was not collected on this outcome measure
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety as Measured by Number of Subjects Who Experience an Adverse Event While on Study Treatment
Time Frame: 6 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 38
Participants | 38

ADVERSE EVENTS:
Time Frame: The average time of Ae collection over all the patient is 6 years
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 11/38
Other Adverse Events (participants affected / at risk) | 31/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=38)
Fever (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Cholangitis (Gastrointestinal disorders) | 1 (1)
Melanoma (Skin and subcutaneous tissue disorders) | 1 (1)
Merkel Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (General disorders) | 2 (2)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Tumor Flare (Blood and lymphatic system disorders) | 2 (2)
Blood Bilirubin Increase (Blood and lymphatic system disorders) | 1 (1)
Infusion Reaction (Injury, poisoning and procedural complications) | 1 (1)
Pruritic Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Shortness of Breath (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=38)
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 23
Neutropenia (Blood and lymphatic system disorders) | 28
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 9
Anemia (Blood and lymphatic system disorders) | 23
Urinary tract Infection (Renal and urinary disorders) | 7
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 15
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial Infection/ Lung Infection (Respiratory, thoracic and mediastinal disorders) | 5
Neutropenic Fever (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 21
Nausea (General disorders) | 12
Vomit (General disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hyperalbuminemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 17
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 13
Hyperglycemia (Metabolism and nutrition disorders) | 19
Elevated Creatinine (Renal and urinary disorders) | 8
Hypertension (Cardiac disorders) | 6
Hypothyroidism (Endocrine disorders) | 6
Hyperthyroidism (Endocrine disorders) | 3
Elevated Alanine Aminotransferase (Hepatobiliary disorders) | 13
Elevated Aspartate Aminotransferase (Hepatobiliary disorders) | 11
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 9
Fever (General disorders) | 22
Fatigue (General disorders) | 28
Night Sweats (General disorders) | 9
Dyspnea (General disorders) | 11
Sore Throat (General disorders) | 9
Cough (General disorders) | 21
Nasal Congestion (Skin and subcutaneous tissue disorders) | 12
Macro Papular (Skin and subcutaneous tissue disorders) | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Cramping (Musculoskeletal and connective tissue disorders) | 6
Gout Flares (Musculoskeletal and connective tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 8
Neuropathy (Nervous system disorders) | 6
Tinnitus (Nervous system disorders) | 5
Abdominal Pain (General disorders) | 9
Head Pain/Headache/Migraine (General disorders) | 10
Rigors (General disorders) | 4
Edema (General disorders) | 16
Chills (General disorders) | 5
Tumor Flare (Blood and lymphatic system disorders) | 13
Infusion Related Reaction (Product Issues) | 13
Serum Sickness (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No